CLINICAL TRIAL: NCT03377335
Title: Effect of Dapagliflozin on Cardio-Metabolic Risk Factors in Patients With Type-2 Diabetes
Brief Title: Dapagliflozin, Cardio-Metabolic Risk Factors and Type-2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Palermo (Other)
Collaborators: AstraZeneca (Industry); University of Catania (Other)
Responsible Party: Principal Investigator, Manfredi Rizzo, Associate Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-16-12388
Record Dates: First submitted 2017-12-09; First posted 2017-12-19 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2017-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Dapagliflozin; Type 2 diabetes mellitus; Carotid intima-media thickness; Endothelial dysfunction; Atherogenic lipoproteins; Inflammatory markers; microRNAs
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin (10mg daily) as add-on to metformin (stable doses ranging from 1500 to 3000 mg daily).
  The total duration of treatment is 6 months.
  Interventions: Drug: Dapagliflozin 10mg
- Metformin alone (Placebo Comparator): Metformin alone (stable doses ranging from 1500 to 3000 mg daily).
  The total duration of treatment is 6 months.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Dapagliflozin 10mg — The subjects in this arm will receive dapagliflozin (10mg daily) as add-on to metformin therapy (doses ranging from 1500 to 3000 mg daily).
  Number of patients to be randomized: 93
  Number of patients expected to complete the study: >87
  All the other medications (including lipid-lowering, anti-hypertensive and anti-platelet agents) will be maintained at fixed doses during the treatment.
  Other Names: Forxiga®
  Arms: Dapagliflozin
Drug: Metformin — All the subjects in this arm will be on metformin therapy only (doses ranging from 1500 to 3000 mg daily).
  Number of patients to be randomized: 93
  Number of patients expected to complete the study: >87
  All the other medications (including lipid-lowering, anti-hypertensive and anti-platelet agents) will be maintained at fixed doses during the treatment.
  Other Names: Glucophage®
  Arms: Metformin alone

SUMMARY:
Dapagliflozin is a member of the sodium-glucose cotransporter-2 (SGLT2) inhibitor class antidiabetes agents which produces significant and sustained reductions in glycemic parameters in patients with type 2 diabetes (T2DM). However, its non-glycemic effects are still largely unknown.

The investigators will evaluate for the first time the effect of dapagliflozin on multiple cardio-metabolic risk markers in one study. So far, no data on the effects of dapagliflozin as well as other SGLT-2 inhibitors on subclinical atherosclerosis, endothelial function, inflammatory markers, cytokines and atherogenic lipoproteins is available.

In addition, the investigators will examine microRNAs (miRNAs) implicated in the development and progression of atherosclerotic disease. Again, no data is currently available on dapaglifozin's as well as other SGLT-2 inhibitors' effects on miRNAs.

The results of this study will show for the first time the potential multiple, non-glycemic effects of dapagliflozin, reducing multiple cardio-metabolic risk markers, which will ultimately lead to decreased CV risk.

In addition, specific mechanisms of the dapagliflozin cardiovascular action will be investigated.

Finally, the results of this study may pave the way for personalized therapy (using the results on miRNAs).

DETAILED DESCRIPTION:
The investigators will perform an open label, two-arms, prospective intervention study using dapagliflozin+metformin vs. metformin alone for a period of 6 months in patients with T2DM.

The research hypothesis is to assess whether dapagliflozin can improve cardio-metabolic outcome, reducing subclinical atherosclerosis, endothelial dysfunction and different cardio-metabolic markers (including inflammatory markers, cytokines, oxidative stress and atherogenic lipoproteins) in patients with T2DM.

The primary objective is to assess the effects of dapagliflozin on subclinical atherosclerosis, as assessed by carotid intima-media thickness (cIMT).

Primary endpoint: Reduction in cIMT.

The secondary objective is to assess the effects of dapagliflozin on glycemic parameters (fasting plasma glucose (FPG), HbA1c), endothelial dysfunction, oxidative stress, atherogenic lipoproteins, inflammatory markers, cytokines and microRNAs (miR-130a, miR-27b, miR-29b and miR-210).

Secondary endpoint: Reduction in glycemic parameters, atherogenic lipoproteins, inflammatory markers, oxidative stress and improvements in endothelial function, cytokines and microRNAs (miR-130a, miR-27b, miR-29b and miR-210).

The full data for clinical and biochemical analyses will be collected in the same fashion at baseline and after 6 months of therapy.

Control visits by the telephone calls will be made every 2 months. However, in case of need, unplanned visits will be scheduled. Unscheduled visits will be performed in case of discontinuation, withdrawal, rescue treatment (including adverse event, episodes of hypoglycemia) or at any time during the study in case of patient's need.

ELIGIBILITY:
Inclusion Criteria:

* men and women with T2DM;
* age >18;
* BMI ≥20 kg/m^2;
* HbA1c 7.0-9.0 %;
* receiving metformin therapy at least 1500 mg/day for at least 8 weeks before screening;
* plasma triglycerides <400 mg/dL, plasma LDL-cholesterol < 250 mg/dL;
* stabile daily dose(s) of hypolipidemic drugs (statins, ezetimibe) for at least 7 weeks prior to the day of randomization;
* adequately controlled blood pressure (≤140/90 mmHg) to be maintained during the study according to Standard of Care;
* able to swallow whole tablets.

Exclusion Criteria:

* pregnancy or willingness to became pregnant;
* severe liver dysfunction (alanine transaminase (ALT) or aspartate transaminase (AST) ≥ 3 times upper limit of normal);
* renal failure with glomerular filtration rate (eGFR) <60 ml/min/1.73m^2;
* major cardiovascular event (myocardial infarction, stroke or hospitalization for unstable angina and/or transient ischaemic attack) within 12 weeks before screening;
* severe infections (such as HIV and HCV);
* any malignancy within 5 years before screening.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2017-12-22 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Subclinical atherosclerosis | Change from baseline to 6 months of the treatment
  To assess the effects of dapagliflozin on subclinical atherosclerosis, as assessed by carotid intima-media thickness (cIMT).

SECONDARY OUTCOMES:
Endothelial dysfunction | Change from baseline to 6 months of the treatment
  To assess the effects of dapagliflozin on endothelial dysfunction through the evaluation of flow mediated dilation (FMD) of the brachial artery.
Oxidative stress | Change from baseline to 6 months of the treatment
  To assess the effects of dapagliflozin on oxidative stress including plasma glutathione, serum lipid hydroperoxides and reactive oxygen species.
Atherogenic lipoproteins | Change from baseline to 6 months of the treatment
  To assess the effects of dapagliflozin on atherogenic lipoproteins including the analysis of the full spectrum of lipoprotein subclasses by gel electrophoresis.
Inflammatory markers | Change from baseline to 6 months of the treatment
  To assess the effects of dapagliflozin on inflammatory markers, including plasma cytokines (pg/ml), that will be assessed using available enzyme-linked immunosorbent assay (ELISA) kits.
microRNAs | Change from baseline to 6 months of the treatment
  To assess the effects of dapagliflozin on microRNAs. The miRNAs are endogenous 21-25 nucleotides noncoding RNA, and they are regulators of gene expression that post transcriptionally modify cellular responses and function. The miRNAs will be isolated from sera using the mirVana miRNA Isolation Kit (Ambion, Waltham, MA, USA), and then quantified by SYBR Green Real-Time (RT) polymerase chain reaction (PCR).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Palermo, Palermo, Italy

REFERENCES:
- [Background] Rizzo M, Rizvi AA, Patti AM, Nikolic D, Giglio RV, Castellino G, Li Volti G, Caprio M, Montalto G, Provenzano V, Genovese S, Ceriello A. Liraglutide improves metabolic parameters and carotid intima-media thickness in diabetic patients with the metabolic syndrome: an 18-month prospective study. Cardiovasc Diabetol. 2016 Dec 3;15(1):162. doi: 10.1186/s12933-016-0480-8. PMID 27912784
- [Background] Rizzo M, Chandalia M, Patti AM, Di Bartolo V, Rizvi AA, Montalto G, Abate N. Liraglutide decreases carotid intima-media thickness in patients with type 2 diabetes: 8-month prospective pilot study. Cardiovasc Diabetol. 2014 Feb 22;13:49. doi: 10.1186/1475-2840-13-49. PMID 24559258
- [Background] Corrado E, Rizzo M, Coppola G, Muratori I, Carella M, Novo S. Endothelial dysfunction and carotid lesions are strong predictors of clinical events in patients with early stages of atherosclerosis: a 24-month follow-up study. Coron Artery Dis. 2008 May;19(3):139-44. doi: 10.1097/MCA.0b013e3282f3fbde. PMID 18418229
- [Background] Salamone F, Galvano F, Marino Gammazza A, Paternostro C, Tibullo D, Bucchieri F, Mangiameli A, Parola M, Bugianesi E, Li Volti G. Silibinin improves hepatic and myocardial injury in mice with nonalcoholic steatohepatitis. Dig Liver Dis. 2012 Apr;44(4):334-42. doi: 10.1016/j.dld.2011.11.010. Epub 2011 Dec 24. PMID 22197629
- [Background] Rizzo M, Abate N, Chandalia M, Rizvi AA, Giglio RV, Nikolic D, Marino Gammazza A, Barbagallo I, Isenovic ER, Banach M, Montalto G, Li Volti G. Liraglutide reduces oxidative stress and restores heme oxygenase-1 and ghrelin levels in patients with type 2 diabetes: a prospective pilot study. J Clin Endocrinol Metab. 2015 Feb;100(2):603-6. doi: 10.1210/jc.2014-2291. Epub 2014 Nov 13. PMID 25393640
- [Background] Berneis K, Rizzo M, Berthold HK, Spinas GA, Krone W, Gouni-Berthold I. Ezetimibe alone or in combination with simvastatin increases small dense low-density lipoproteins in healthy men: a randomized trial. Eur Heart J. 2010 Jul;31(13):1633-9. doi: 10.1093/eurheartj/ehq181. Epub 2010 Jun 6. PMID 20525999
- [Background] Mikhailidis DP, Elisaf M, Rizzo M, Berneis K, Griffin B, Zambon A, Athyros V, de Graaf J, Marz W, Parhofer KG, Rini GB, Spinas GA, Tomkin GH, Tselepis AD, Wierzbicki AS, Winkler K, Florentin M, Liberopoulos E. "European panel on low density lipoprotein (LDL) subclasses": a statement on the pathophysiology, atherogenicity and clinical significance of LDL subclasses. Curr Vasc Pharmacol. 2011 Sep;9(5):533-71. doi: 10.2174/157016111796642661. PMID 21595628
- [Background] Barbagallo I, Parenti R, Zappala A, Vanella L, Tibullo D, Pepe F, Onni T, Li Volti G. Combined inhibition of Hsp90 and heme oxygenase-1 induces apoptosis and endoplasmic reticulum stress in melanoma. Acta Histochem. 2015 Oct;117(8):705-11. doi: 10.1016/j.acthis.2015.09.005. Epub 2015 Oct 19. PMID 26493719
- [Background] Cengiz M, Yavuzer S, Kilickiran Avci B, Yuruyen M, Yavuzer H, Dikici SA, Karatas OF, Ozen M, Uzun H, Ongen Z. Circulating miR-21 and eNOS in subclinical atherosclerosis in patients with hypertension. Clin Exp Hypertens. 2015;37(8):643-9. doi: 10.3109/10641963.2015.1036064. Epub 2015 Jun 26. PMID 26114349
- [Background] Tziomalos K, Athyros VG, Karagiannis A. Editorial: Vascular Calcification, Cardiovascular Risk and microRNAs. Curr Vasc Pharmacol. 2016;14(2):208-10. doi: 10.2174/157016111402160208150816. PMID 26864445
- [Background] Signorelli SS, Volsi GL, Pitruzzella A, Fiore V, Mangiafico M, Vanella L, Parenti R, Rizzo M, Volti GL. Circulating miR-130a, miR-27b, and miR-210 in Patients With Peripheral Artery Disease and Their Potential Relationship With Oxidative Stress. Angiology. 2016 Nov;67(10):945-950. doi: 10.1177/0003319716638242. Epub 2016 Jul 11. PMID 26980776
- [Background] Peng H, Zhong M, Zhao W, Wang C, Zhang J, Liu X, Li Y, Paudel SD, Wang Q, Lou T. Urinary miR-29 correlates with albuminuria and carotid intima-media thickness in type 2 diabetes patients. PLoS One. 2013 Dec 9;8(12):e82607. doi: 10.1371/journal.pone.0082607. eCollection 2013. PMID 24349318